CLINICAL TRIAL: NCT01218659
Title: A Randomized, Open-Label Study to Compare the Efficacy and Safety of AT1001 and Enzyme Replacement Therapy (ERT) in Patients With Fabry Disease and AT1001-Responsive GLA Mutations, Who Were Previously Treated With ERT
Brief Title: Study to Compare the Efficacy and Safety of Oral AT1001 and Enzyme Replacement Therapy in Patients With Fabry Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT1001-012; ATTRACT (Other: Amicus Therapeutics); 2010-022636-37 (EudraCT Number)
Record Dates: First submitted 2010-10-06; First posted 2010-10-11 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Fabry Disease
Keywords: Amicus Therapeutics; Galafold; AT1001; Migalastat
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate; agalsidase beta; agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Migalastat (Experimental): Participants received 150 mg migalastat orally QOD during the 18-month randomized treatment period and the optional 12-month OLE period. Participants received an inactive reminder capsule on alternate days during both treatment periods.
  Interventions: Drug: migalastat hydrochloride
- ERT (Active Comparator): Participants received ERT (either agalsidase alfa or agalsidase beta) as prescribed by the participant's treating physician and administered in accordance with the approved prescribing information during the 18-month randomized treatment period. Participants were required to be given >80% of the currently labeled dose and regimen during the 18-month randomized treatment period. During the optional 12-month OLE period, participants received 150 mg migalastat orally QOD. Participants received an inactive reminder capsule on alternate days during the OLE.
  Interventions: Biological: agalsidase

INTERVENTIONS:
Drug: migalastat hydrochloride — 150-mg capsule administered orally QOD
  Other Names: AT1001; Migalastat; Galafold
  Arms: Migalastat
Biological: agalsidase — Agalsidase via intravenous infusion as prescribed by the participant's treating physician and in accordance with the approved prescribing information
  Other Names: agalsidase beta; Fabrazyme; agalsidase alfa; Replagal
  Arms: ERT

SUMMARY:
Study to compare the efficacy and safety of migalastat and enzyme replacement therapy (ERT) in male and female participants with Fabry disease who are currently receiving ERT and who have an alpha galactosidase-A (α Gal-A) mutation that is amenable to migalastat, based on the clinical trial human embryonic kidney cell (HEK) assay.

DETAILED DESCRIPTION:
This was a Phase 3, randomized, open-label, active-controlled study to evaluate the efficacy and safety of 150 milligrams (mg) of migalastat hydrochloride (migalastat) (equivalent to 123 mg of migalastat) once every other day (QOD) and ERT in male and female participants with Fabry disease who were receiving ERT and who have an α Gal-A mutation that is amenable to migalastat, based on the clinical trial HEK assay. This was a 2-part study. Part 1, the 18-month randomized phase, evaluated participants who received either migalastat 150 mg QOD or ERT per prescribing physicians' instructions for efficacy and safety. Part 2, the optional 12-month open-label extension (OLE) phase in which all participants received migalastat, also explored efficacy and safety. For Part 2, all participants who received ERT in Part 1 were given migalastat. Data presented in this posting include efficacy data from the 18-month randomized period and safety data from the entire study (18-month randomized period and 12-month optional OLE [total of 30 months]).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 16 and 74 diagnosed with Fabry disease
* Confirmed α Gal-A mutation that is amenable to migalastat, based on the clinical trial HEK assay
* Participant has been on ERT for at least 12 months before screening/baseline
* Dose level and regimen of ERT have been stable for 3 months before screening/baseline and is at least 80% of the currently labeled dose and regimen for this time period
* Glomerular filtration rate (GFR) ≥ 30 milliliter (mL)/minute (min) /1.73 m^2
* Participants taking angiotensin converting enzyme inhibitors or angiotensin receptor blockers must be on a stable dose for at least 4 weeks before screening/baseline
* Women who can become pregnant and all men agree to be sexually abstinent or use medically accepted methods of birth control throughout the duration of the study and for up to 30 days after last dose of study medication
* Participant is willing and able to provide written informed consent and assent if applicable

Exclusion Criteria:

* Participant has undergone, or is scheduled to undergo, kidney transplantation or any other solid organ transplantation
* Participant is on regular dialysis that is specifically for the treatment of chronic kidney disease
* Participant has had a documented transient ischemic attack, stroke, unstable angina, or myocardial infarction within the 3 months before screening/baseline
* Participant has clinically significant unstable cardiac disease in the opinion of the investigator (for example, cardiac disease requiring active management, such as symptomatic arrhythmia, unstable angina, or New York Heart Association (NYHA) class III or IV congestive heart failure)
* Pregnant or breast-feeding
* History of allergy or sensitivity to study medication (including excipients) or other iminosugars (for example, miglustat, miglitol)
* Participant has absolute contraindication to iohexol and/or inability to undergo iohexol GFR testing
* Participant requires treatment with Glyset® (miglitol), or Zavesca® (miglustat)
* Participant received any investigational/experimental drug, biologic or device within 30 days of screening/baseline
* Any intercurrent illness or condition that may preclude the participant from fulfilling the study requirements or suggests to the investigator that the participant may have an unacceptable risk by participating in this study

Ages: 16 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-09-08 (Actual); Primary Completion 2014-05-27 (Actual); Study Completion 2015-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (23):
- United States (8):
  - Los Angeles, California
  - Aurora, Colorado
  - Decatur, Georgia
  - Grand Rapids, Michigan
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Fairfax, Virginia
  - Milwaukee, Wisconsin
- Australia (2):
  - Parkville, Victoria
  - Perth, Western Australia
- Vienna, Austria
- Edegem, Belgium
- São Paulo, Brazil
- Copenhagen, Denmark
- France (2):
  - Garches
  - Lille
- Florence, Italy
- Japan (3):
  - Niigata
  - Osaka
  - Tokyo
- United Kingdom (3):
  - Cambridge
  - London
  - Salford

REFERENCES:
- [Derived] Feldt-Rasmussen U, Hughes D, Sunder-Plassmann G, Shankar S, Nedd K, Olivotto I, Ortiz D, Ohashi T, Hamazaki T, Skuban N, Yu J, Barth JA, Nicholls K. Long-term efficacy and safety of migalastat treatment in Fabry disease: 30-month results from the open-label extension of the randomized, phase 3 ATTRACT study. Mol Genet Metab. 2020 Sep-Oct;131(1-2):219-228. doi: 10.1016/j.ymgme.2020.07.007. Epub 2020 Aug 15. PMID 33012654
- [Derived] Bichet DG, Aerts JM, Auray-Blais C, Maruyama H, Mehta AB, Skuban N, Krusinska E, Schiffmann R. Assessment of plasma lyso-Gb3 for clinical monitoring of treatment response in migalastat-treated patients with Fabry disease. Genet Med. 2021 Jan;23(1):192-201. doi: 10.1038/s41436-020-00968-z. Epub 2020 Sep 30. PMID 32994552
- [Derived] Haninger-Vacariu N, El-Hadi S, Pauler U, Foretnik M, Kain R, Prohaszka Z, Schmidt A, Skuban N, Barth JA, Sunder-Plassmann G. Pregnancy Outcome after Exposure to Migalastat for Fabry Disease: A Clinical Report. Case Rep Obstet Gynecol. 2019 Dec 21;2019:1030259. doi: 10.1155/2019/1030259. eCollection 2019. PMID 31934472
- [Derived] Narita I, Ohashi T, Sakai N, Hamazaki T, Skuban N, Castelli JP, Lagast H, Barth JA. Efficacy and safety of migalastat in a Japanese population: a subgroup analysis of the ATTRACT study. Clin Exp Nephrol. 2020 Feb;24(2):157-166. doi: 10.1007/s10157-019-01810-w. Epub 2019 Dec 30. PMID 31889231
- [Derived] Hughes DA, Nicholls K, Shankar SP, Sunder-Plassmann G, Koeller D, Nedd K, Vockley G, Hamazaki T, Lachmann R, Ohashi T, Olivotto I, Sakai N, Deegan P, Dimmock D, Eyskens F, Germain DP, Goker-Alpan O, Hachulla E, Jovanovic A, Lourenco CM, Narita I, Thomas M, Wilcox WR, Bichet DG, Schiffmann R, Ludington E, Viereck C, Kirk J, Yu J, Johnson F, Boudes P, Benjamin ER, Lockhart DJ, Barlow C, Skuban N, Castelli JP, Barth J, Feldt-Rasmussen U. Oral pharmacological chaperone migalastat compared with enzyme replacement therapy in Fabry disease: 18-month results from the randomised phase III ATTRACT study. J Med Genet. 2017 Apr;54(4):288-296. doi: 10.1136/jmedgenet-2016-104178. Epub 2016 Nov 10. PMID 27834756
- [Derived] Benjamin ER, Della Valle MC, Wu X, Katz E, Pruthi F, Bond S, Bronfin B, Williams H, Yu J, Bichet DG, Germain DP, Giugliani R, Hughes D, Schiffmann R, Wilcox WR, Desnick RJ, Kirk J, Barth J, Barlow C, Valenzano KJ, Castelli J, Lockhart DJ. The validation of pharmacogenetics for the identification of Fabry patients to be treated with migalastat. Genet Med. 2017 Apr;19(4):430-438. doi: 10.1038/gim.2016.122. Epub 2016 Sep 22. PMID 27657681

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The All Migalastat group was comprised of participants who received migalastat during the randomized treatment period (0-18 mo.) and who received enzyme replacement therapy (ERT) during the randomized treatment period (0-18 mo.) and switched to migalastat during the 12-mo. open-label extension (OLE). 8 participants enrolled but did not randomize.
Groups:
- Migalastat (0-18 Months): Participants received 150 milligrams (mg) of migalastat hydrochloride (migalastat) (equivalent to 123 mg of migalastat) orally once every other day (QOD) during the 18-month randomized treatment period (0-18 months). Participants received an inactive reminder capsule on alternate days during both treatment periods.
- ERT (0-18 Months): Participants received ERT (either agalsidase alfa or agalsidase beta) as prescribed by the participant's treating physician and administered in accordance with the approved prescribing information during the 18-month randomized treatment period (0-18 months). Participants were required to be given >80% of the currently labeled dose and regimen during the 18-month randomized treatment period.
- All Migalastat (0-30 Months): Participants in this group are composed of participants from the Migalastat (0-18 months) and the ERT (0-18 months) groups. Therefore, participants in the All Migalastat group received at least 1 dose of 150 mg migalastat orally QOD during the 18-month randomization period or the optional 12-month OLE (for a total time period of up to 30 months), regardless of whether or not the participant discontinued the study early, and regardless of whether they were previously randomized to migalastat or ERT during the 18-month Randomized Period (0-18 months).
Period: 18-Month Randomized Period
Arm/Group | Migalastat (0-18 Months) | ERT (0-18 Months) | All Migalastat (0-30 Months)
Started | 36 | 24 | 0 (Zero participants are noted here because participants started in this group during the 12-month OLE.)
Safety Population (Safety: received at least 1 dose of migalastat or ERT.) | 36 | 21 | 0 (Zero participants are noted here because participants started in this group during the 12-month OLE.)
Completed | 34 | 18 | 0 (Zero participants are noted here because participants started in this group during the 12-month OLE.)
Not Completed | 2 | 6 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0
Not completed — Did not receive study drug | 0 | 3 | 0
Period: 12-Month OLE
Arm/Group | Migalastat (0-18 Months) | ERT (0-18 Months) | All Migalastat (0-30 Months)
Started | 0 (Zero participants are noted here because they were combined in the All Migalastat (0-30 mo.) group.) | 0 (Zero participants are noted here because they were combined in the All Migalastat (0-30 mo.) group.) | 52 (Fifty-two participants completed the 18-mo. randomized treatment period.)
Safety Population (Safety: ITT pop. who received ≥1 dose of study drug during the 18-mo randomized treatment period.) | 0 | 0 | 51
Modified Intent-to-Treat (mITT) (mITT: Eligibility based on Good Laboratory Practice (GLP) human embryonic kidney cell (HEK) assay.) | 0 (Zero participants are noted here because they were combined in the All Migalastat (0-30 mo.) group.) | 0 (Zero participants are noted here because they were combined in the All Migalastat (0-30 mo.) group.) | 46
Completed | 0 (Zero participants are noted here because they were combined in the All Migalastat (0-30 mo.) group.) | 0 (Zero participants are noted here because they were combined in the All Migalastat (0-30 mo.) group.) | 42
Not Completed | 0 | 0 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Declined to participate in the OLE | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Safety Population: All randomized participants who received at least 1 dose of migalastat or ERT.
Groups:
- Migalastat (0-18 Months): Participants received 150 mg migalastat orally QOD during the 18-month randomized treatment period. Participants received an inactive reminder capsule on alternate days during both treatment periods.
- ERT (0-18 Months): Participants received ERT (either agalsidase alfa or agalsidase beta) as prescribed by the participant's treating physician and administered in accordance with the approved prescribing information during the 18-month randomized treatment period. Participants were required to be given >80% of the currently labeled dose and regimen during the 18-month randomized treatment period. Participants received an inactive reminder capsule on alternate days during the OLE.
- Total: Total of all reporting groups
Arm/Group | Migalastat (0-18 Months) | ERT (0-18 Months) | Total
Number analyzed (Participants) | 36 | 21 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (13.76) | 46.3 (14.91) | 48.9 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 16 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate Of Change From Baseline To Month 18 In Measured Glomerular Filtration Rate
Description: To assess renal function, measured glomerular filtration rate (GFR) was measured by the plasma clearance of unlabeled iohexol (mGFR-iohexol), a non-ionic contrast agent. The annualized rate of change in mGFR-iohexol from Baseline to Month 18 was analyzed using an analysis of covariance (ANCOVA) model with the following factors as covariates: treatment group, sex, age, Baseline GFR (mGFR-iohexol), and Baseline 24-hour (hr) urine protein. A threshold of <2.2 milliliter (mL)/minute (min)/1.73 meter squared (m^2)/year was established to compare migalastat to ERT. This difference of 2.2 mL/min/1.73 m2/year is based on the smallest expected rate of decline in estimated glomerular filtration rate (eGFR) for participants treated with agalsidase alfa for 18 months.
Time Frame: Baseline to Month 18
Population: mITT Population: All randomized participants with an α Gal-A mutation that is amenable to migalastat, based on the GLP HEK assay, who received at least 1 dose of study drug, had Baseline and postbaseline mGFR-iohexol values, and postbaseline measure of the estimated GFR using the CKD-EPI equation.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2/year
Groups:
- ERT (0-18 Months): Participants received ERT (either agalsidase alfa or agalsidase beta) as prescribed by the participant's treating physician and administered in accordance with the approved prescribing information during the 18-month randomized treatment period. Participants were required to be given >80% of the currently labeled dose and regimen during the 18-month randomized treatment period. During the optional 12-month OLE period, participants received 150 mg migalastat orally QOD. Participants received an inactive reminder capsule on alternate days during the OLE.
Arm/Group | Migalastat (0-18 Months) | ERT (0-18 Months)
Number analyzed (Participants) | 34 | 18
mL/min/1.73 m^2/year | -4.35 [-7.65 to -1.06] | -3.24 [-7.81 to 1.33]

2. Primary Outcome: Annualized Rate Of Change From Baseline To Month 18 In eGFR
Description: The eGFR assessed by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation was calculated using the following:
  eGFR-CKD-EPI = 141 x min (Serum Creatinine/κ,1)^(α) x max(Serum Creatinine/κ,1)^(-1.209) x 0.993^(Age) x 1.1018 (if female) x 1.159 (if African American or black) where: κ is 0.7 for females and 0.9 for males; α is -0.329 for females and -0.411 for males; min indicates the minimum of Serum Creatinine/κ or 1; max indicates the maximum of Serum Creatinine/κ or 1.
  The annualized rate of change in eGFR-CKD-EPI from Baseline to Month 18 was analyzed using an ANCOVA model with the following factors as covariates: treatment group, sex, age, Baseline GFR (eGFR-CKD-EPI), and Baseline 24-hr urine protein. A threshold of <2.2 mL/min/1.73m^2/year was established to compare migalastat to ERT. This difference of 2.2 mL/min/1.73 m2/year is based on the smallest expected rate of decline in eGFR for participants treated with agalsidase alfa for 18 months.
Time Frame: Baseline to Month 18
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2/year
Arm/Group | Migalastat (0-18 Months) | ERT (0-18 Months)
Number analyzed (Participants) | 34 | 18
mL/min/1.73 m^2/year | -0.40 [-2.27 to 1.48] | -1.03 [-3.64 to 1.58]

3. Secondary Outcome: Annualized Rate Of Change From Baseline To Month 18 In eGFR By The Modification Of Diet In Renal Disease Equation
Description: The GFR estimated by the Modification Of Diet In Renal Disease equation (eGFR-MDRD) was calculated using the following equation: eGFR-MDRD = 175 x (Serum Creatinine)^(-1.154) x (Age)^(-0.203) x 1.212 (if participant's race is black or African American) x 0.742 (if participant is female).
  The eGFR-MDRD from Baseline to Month 18 was analyzed using an ANCOVA model with the following factors as covariates: treatment group, sex, age, Baseline GFR (eGFR-CKD-EPI), and Baseline 24-hr urine protein.
Time Frame: Baseline to Month 18
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2/year
Arm/Group | Migalastat (0-18 Months) | ERT (0-18 Months)
Number analyzed (Participants) | 34 | 18
mL/min/1.73 m^2/year | -1.51 [-3.43 to 0.40] | -1.53 [-4.20 to 1.13]

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data were collected from the time of signing informed consent at screening/baseline through the follow-up visit (1 mo. after the last treatment in the optional OLE/after the 18-month Randomized Period if the participant did not enroll in the OLE), for up to 30 months. Because participants in the Migalastat (0-18 mo.) and ERT (0-18 mo.) groups were combined into the All Migalastat (0-30 mo.) group, AEs for those groups are included in the All Migalastat (0-30 mo.) group AEs.
Groups:
- Migalastat (0-18 Months): Participants received 150 mg of migalastat orally QOD during the 18-month randomized treatment period (0-18 months). Participants received an inactive reminder capsule on alternate days during both treatment periods.
- All Migalastat (0-30 Months): Participants in this group are composed of participants from the Migalastat (0-18 month) and the ERT (0-18 month) groups. Therefore, participants in the All Migalastat group received at least 1 dose of 150 mg migalastat orally QOD during the 18-month randomized treatment period or the optional 12-month OLE (for a total time period of up to 30 months), regardless of whether or not the participant discontinued the study early, and regardless of whether they were previously randomized to migalastat or ERT during the 18-month randomized phase (0-18 months).
Arm/Group | Migalastat (0-18 Months) | ERT (0-18 Months) | All Migalastat (0-30 Months)
Serious Adverse Events (participants affected / at risk) | 7/36 | 7/21 | 16/51
Other Adverse Events (participants affected / at risk) | 34/36 | 20/21 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (0-18 Months) (N=36) | ERT (0-18 Months) (N=21) | All Migalastat (0-30 Months) (N=51)
Pneumonia (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1
Perineal abscess (Infections and infestations) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 1 | 2
Chest pain (General disorders) | 3 | 0 | 3
Device malfunction (General disorders) | 0 | 1 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (0-18 Months) (N=36) | ERT (0-18 Months) (N=21) | All Migalastat (0-30 Months) (N=51)
Palpitations (Cardiac disorders) | 2 | 1 | 5
Tinnitus (Ear and labyrinth disorders) | 3 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 11
Nausea (Gastrointestinal disorders) | 5 | 2 | 8
Vomiting (Gastrointestinal disorders) | 3 | 3 | 8
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 7
Constipation (Gastrointestinal disorders) | 3 | 1 | 4
Toothache (Gastrointestinal disorders) | 3 | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 3
Flatulence (Gastrointestinal disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 3 | 1 | 6
Influenza like illness (General disorders) | 2 | 0 | 3
Oedema peripheral (General disorders) | 2 | 2 | 2
Nasopharyngitis (Infections and infestations) | 12 | 7 | 21
Influenza (Infections and infestations) | 5 | 4 | 12
Urinary tract infection (Infections and infestations) | 4 | 1 | 6
Bronchitis (Infections and infestations) | 2 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 5
Sinusitis (Infections and infestations) | 3 | 3 | 4
Herpes Zoster (Infections and infestations) | 2 | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 3
Gastroenteritis (Infections and infestations) | 2 | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 4
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 7
Protein urine present (Investigations) | 3 | 0 | 4
White blood cell count decreased (Investigations) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Headache (Nervous system disorders) | 9 | 5 | 16
Dizziness (Nervous system disorders) | 6 | 2 | 8
Presyncope (Nervous system disorders) | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0 | 5
Depression (Psychiatric disorders) | 2 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Cystitis (Infections and infestations) | 1 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Neuralgia (Nervous system disorders) | 1 | 1 | 4
Paraesthesia (Nervous system disorders) | 1 | 0 | 3
Tremor (Nervous system disorders) | 1 | 0 | 3
Pain (General disorders) | 1 | 0 | 5
Fatigue (General disorders) | 1 | 1 | 4
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results from this trial, provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review prior to submission for publication. If requested and prior to publication, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.